CLINICAL TRIAL: NCT01244022
Title: Postoperative Serum Cytokine Changes After Radical Resection of Colorectal Cancer
Brief Title: Cytokine Changes After Colorectal Cancer Resection
Status: Completed | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Drazen Servis, M.D., Ph. D., University Hospital Dubrava
Other Study IDs: DS-P03112010
Record Dates: First submitted 2010-11-12; First posted 2010-11-19 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Surgical stress response; interleukins
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each patient, serum samples will be stored at -80°C for later determining of serum cytokine levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Patients with pathohistologically verified colorectal cancer or adenoma with epithelial dysplasia
  Interventions: Procedure: colorectal cancer resection

INTERVENTIONS:
Procedure: colorectal cancer resection — Open radical resection of colorectal cancer, according to oncological principals, depending on the tumor site
  Other Names: Hemicolectomy; Rectosigmoid resection

SUMMARY:
Based on our previous research, this study aims to determine reliable surgical stress response markers in patients undergoing radical resection of colorectal cancer.

DETAILED DESCRIPTION:
Every surgical intervention represents a stress for patient's organism. During the operation, numerous changes in the patient's metabolism take place, that are termed surgical stress response. Leading cause of surgical stress response is tissue destruction that always accompanies operations. Surgical stress response is effected through activation of hypothalamus-pituitary-adrenal axis and through sympathetic activation.

The consequences of surgical stress response are numerous. Surgical stress response is essential to uneventful postoperative recovery. On the other hand, excessive surgical stress response may lead to serious postoperative complications, such as heart and kidney failure, venous thrombosis, disruption of operative wound and wound infection.

In prior studies the investigators have shown the kinetics of postoperative serum interleukin changes after radical resection of gastric cancer.

This study aims at determining reliable markers of surgical stress response severity in patients undergoing radical resection of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathohistologically verified colorectal cancer

Exclusion Criteria:

* Distant metastases noticed before or during surgery
* History of autoimmune diseases or immunodeficiencies
* Use of immunomodulatory drugs within 1 year prior to surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer treated in the University Hospital Dubrava
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postoperative changes of serum cytokine levels | 1 day, 2 days and 7 days postoperatively
  Serum cytokine levels will be determined at 1st, 2nd and 7th postoperative day and compared to preoperative values.

SECONDARY OUTCOMES:
Early postoperative complications | Within one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Drazen Servis, M.D., Ph.D., Principal Investigator — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Background] Servis D, Busic Z, Stipancic I, Patrlj L, Gagro A. Serum cytokine changes after gastric resection or gastrectomy for gastric cancer. Hepatogastroenterology. 2008 Sep-Oct;55(86-87):1868-72. PMID 19102411
- [Derived] Etherek L, Servis D, Unic A. Soluble Triggering Receptor Expressed on Myeloid Cells-1 and Inflammatory Markers in Colorectal Cancer Surgery: A Prospective Cohort Study. Chin Med J (Engl). 2017 Nov 20;130(22):2691-2696. doi: 10.4103/0366-6999.218022. PMID 29133757